CLINICAL TRIAL: NCT03606655
Title: A Single-Arm Pre- and Post-Pilot Trial Exploring the Impact of Two-week Kava on the Metabolism of Two Tobacco Chemicals, Nicotine and NNK, in Head and Neck Cancer Survivors Who Are Active Smokers
Brief Title: Exploring the Impact of Two-week Kava on the Metabolism of Nicotine and NNK
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Terms could not be met with the FDA.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB201801361; UF-PDO-HN-1001 (Other: University of Florida); OCR18359 (Other: University of Florida)
Record Dates: First submitted 2018-07-20; First posted 2018-07-31 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Kava on the Metabolism of Nicotine and NNK
Keywords: kava; tobacco; cessation; cancer; nicotine; NNK; metabolism; carcinogen
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Single-Arm Pre- and Post- Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Kava (Experimental): This is a single-arm pre- and post- Phase 0/1 study with one primary goal to explore the feasibility of recruitment of participants, adherence rate, acceptability of treatment and completion rate with 14 day dietary supplement kava treatment in head and neck cancer patients who continue to smoke. The other primary goal is to evaluate distribution of change in nicotine and NNK metabolism after 14 day kava treatment..
  Interventions: Drug: Kava

INTERVENTIONS:
Drug: Kava — Kava: 75 mg three times daily (3 capsules)

SUMMARY:
Tobacco smoking is the leading cause of head and neck cancer in the United States. Smoking cessation remains a challenge for many head/neck cancer survivors, indicating a need for development of more effective smoking cessation interventions. Kava's properties as a proven anxiolytic and carcinogen detoxifier warrant an investigation of its efficacy as an innovative smoking cessation aid. Kava may also influence carcinogen (NNK specifically) metabolism to help reduce carcinogenesis risk.

DETAILED DESCRIPTION:
Tobacco smoking is the leading cause of head and neck cancer in the United States and a significant portion of head/neck cancer survivors continue to smoke even though smoking negatively impacts their clinical outcomes and increases chance of recurrence. Two tobacco chemicals, NNK and nicotine, are respectively responsible for the increased recurrence risk and tobacco addiction. Kava s properties as a proven anxiolytic and a potential carcinogen detoxifier warrant an investigation of its effects on the metabolism of these two tobacco chemicals among head/neck cancer survivors who continue to smoke. The results will identifying surrogate biomarkers and provide information regarding kava s potential as a future intervention to both promote smoking cessation and reduce carcinogenesis risk.

Primary Objective:

To explore the feasibility of recruitment of participants, adherence rate, acceptability of treatment and completion rate with 14 day dietary supplement kava treatment in head and neck cancer patients who continue to smoke.

To evaluate distribution of change in nicotine and NNK metabolism after 14 day kava treatment.

Exploratory Objective:

To evaluate distribution of change in mood after 14 day kava treatment. To evaluate prevalence of pain and pain medication use and distribution of change in pain and pain medication consumption after 14 day kava treatment.

ELIGIBILITY:
Inclusion Criteria:

Individuals eligible for study participation must meet the following criteria:

* Must be a current smoker with history of head and neck cancer.
* Must be at least 3 months out from completing definitive cancer treatment.
* Must not be undergoing active treatment for cancer or have known recurrence.
* Subjects must have adequate organ function, as defined by: the clinical chemistry analysis of ALT, ALP, AST and total bilirubin within the normal range.
* Subjects must have access to a functional telephone.
* Written informed consent obtained from the subject or the subject's legal representative and the ability for the subject to comply with all the study-related procedures.
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study. Prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.

WOCBP include any woman who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or who is not post-menopausal. Post-menopause is defined as:

* Amenorrhea that has lasted for ≥ 12 consecutive months without another cause, or
* For women with irregular menstrual periods who are taking hormone replacement therapy (HRT), a documented serum follicle-stimulating hormone (FSH) level of greater than 35 mIU/mL.
* Males with female partners of child-bearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study.

Exclusion Criteria:

Subjects with any of the following will not be eligible for study participation:

* Known liver disease as defined by the following elevated serum levels of AST, ALK Phos, ALT or total bilirubin:
* Consumption of more than three alcoholic drinks per day
* D. Subjects must not have been diagnosed with any liver dysfunction
* Subjects who regularly take more than the recommended dose of acetaminophen for pain management.
* Females or males of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period.
* Females who are pregnant or breastfeeding.
* History of any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician.
* Prisoners or subjects who are involuntarily incarcerated.
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.
* Subjects demonstrating an inability to comply with the study and/or follow-up procedures.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Total NNAL | Two weeks
  Total NNAL (the creatinine-normalized sum of NNAL, NNAL-N-gluc, and NNAL-O-gluc) will be calculated via urinary analysis at the screening visit and the final study visit to determine kava's effect on the pharmacokinetics and metabolism of carcinogens [NNK: 4-(methylnitrosamino)-1-3(pyridyl)-1-butanone].
The ratio of total NNAL-gluc to NNAL | Two weeks
  The ratio of total NNAL-gluc to NNAL will be calculated via urinary analysis at the screening visit and the final study visit to determine kava's effect on the pharmacokinetics and metabolism of carcinogens [NNK: 4-(methylnitrosamino)-1-3(pyridyl)-1-butanone].
The urinary DNA adducts of 3-mA upon TNE correction | Two weeks
  The urinary DNA adducts of 3-mA upon TNE correction will be calculated via urinary analysis at the screening visit and the final study visit to determine kava's effect on the pharmacokinetics and metabolism of carcinogens [NNK: 4-(methylnitrosamino)-1-3(pyridyl)-1-butanone].
The ratio of total NNAL to TNE | Two weeks
  The ratio of total NNAL to TNE (the creatinine-normalized sum of total nicotine, total cotinine, total 3-hydroxycotinine, and nicotine N-oxide) will be calculated via urinary analysis at the screening visit and the final study visit to determine kava's effect on the pharmacokinetics and metabolism of carcinogens [NNK: 4-(methylnitrosamino)-1-3(pyridyl)-1-butanone].
The DNA adducts in the buccal cells from oral swab | Two weeks
  The DNA adducts in the buccal cells will be calculated via oral swab at the screening visit and the final study visit to determine kava's effect on the pharmacokinetics and metabolism of carcinogens [NNK: 4-(methylnitrosamino)-1-3(pyridyl)-1-butanone].

SECONDARY OUTCOMES:
Positive and Negative Affect Scale (PANAS) | Two weeks
  The efficacy of the dietary supplement kava to positively affect mood will be evaluated via questionnaire. The PANAS scale consists of 20 words that describe different feelings and emotions that can be rated as: 1) Very slightly or not at all 2) A little 3) Moderately 4) Quite a bit 5) Extremely. This questionnaire will be completed at the initial study visit and at the final study visit.
WHO Quality of Life BREF (WHOQOL-BREF) | Two weeks
  Kava's effect on pain and pain medicine consumption will be evaluated via questionnaire. The WHOQOL-BREF instrument comprises 26 items, which measure the following broad domains: physical health, psychological health, social relationships, and environment. This questionnaire will be completed at the initial study visit and at the final study visit.
Brief Pain Inventory Questionnaire | Two weeks
  Kava's effect on pain and pain medicine consumption will be evaluated via questionnaire. The purpose of the BPI is to assess the severity of pain and the impact of pain on daily functions, and focuses on patients with pain from chronic diseases or conditions such as cancer, osteoarthritis and low back pain, or with pain from acute conditions such as postoperative pain. It assesses areas of pain severity, impact of pain on daily function, location of pain, pain medications and amount of pain relief in the past 24 hours or the past week. This questionnaire will be completed at the initial study visit and at the final study visit.

OTHER OUTCOMES:
Minnesota Nicotine Withdrawal Scale (MNWS) | Two weeks
  The efficacy of the dietary supplement kava to reduce tobacco use will be evaluated via questionnaire. The MNWS is used to assess withdrawal symptoms. The nine items of the MNWS included the following: urge to smoke (craving); depressed mood; irritability, frustration, or anger; anxiety; difficulty concentrating; restlessness; increased appetite; difficulty going to sleep; and difficulty staying asleep. Each item was rated by a subject on an ordinal scale from 0 (not at all) to 4 (extreme). This questionnaire will be completed at the initial study visit and at the final study visit.
Fagerstrom Test Nicotine Dependence (FTND) | Two weeks
  The efficacy of the dietary supplement kava to reduce tobacco use will be evaluated via questionnaire. The FTND is a standard instrument for assessing the intensity of physical addiction to nicotine. This test was designed to provide an ordinal measure of nicotine dependence related to cigarette smoking. It contains six items that evaluate the quantity of cigarette consumption, the compulsion to use, and dependence. This questionnaire will be completed at the initial study visit and at the final study visit.
Brief Questionnaire of Smoking Urges (QSU-Brief) | Two weeks
  The efficacy of the dietary supplement kava to reduce tobacco use will be evaluated via questionnaire. The QSU-Brief questionnaire consists of 10 items comprising four putative features of craving including anticipation of relief of nicotine withdrawal, anticipation of positive outcomes of smoking, desire to smoke, and intention to smoke. This questionnaire will be completed at the initial study visit and at the final study visit.
Modified Cigarette Evaluation Scale (mCES) | Two weeks
  The efficacy of the dietary supplement kava to reduce tobacco use will be evaluated via questionnaire. The mCES contains 12 items rated on a 0-6 point Likert scale from 'not at all' to 'extremely'. The mCES is comprised of several subscales: Smoking Satisfaction, Psychological Reward, Aversion, Enjoyment of Respiratory Tract Sensations, and Craving Reduction. This questionnaire will be completed at the initial study visit and at the final study visit.
Cancer Patient Tobacco Use Questionnaire (C-TUQ) | Two weeks
  The efficacy of the dietary supplement kava to reduce tobacco use will be evaluated via questionnaire. The C-TUQ is a 22-item self-report survey designed to capture information about tobacco use by cancer patients and cancer survivors. The C-TUQ survey tool is divided into five domains: 1) Basic Tobacco Use Information 2) Cigarette Smoking in Relation to Cancer Diagnosis and Treatment 3) Smoking Cessation, Cessation Products, and Assistance Methods 4) Use of Other Products 5) Second-Hand Smoke Exposure. This questionnaire will be completed at the initial study visit and at the final study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Silver, MD, Principal Investigator — University of Florida

IPD SHARING:
Plan to Share IPD: No